CLINICAL TRIAL: NCT02557932
Title: Comparison of 7-day Proton Pump Inhibitor (PPI)-Clarithromycin Containing Triple Therapy and 10-day Bismuth Quadruple Therapy for Helicobacter Eradication as First-line Regimen: Randomized Controlled Trial
Brief Title: Comparison of 7-day PPI-based Standard Triple Therapy and 10-day Bismuth Quadruple Therapy for H. Pylori Eradication
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Il Ju Choi, Department of gastroenterology, Center for Gastric Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2015-0207
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Helicobacter Pylori Infection; Family History of Stomach Cancer
Keywords: PPI standard triple therapy; Bismuth quadruple therapy; Helicobacter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard triple therapy (Active Comparator): 7 day-PPI based standard triple therapy
  Interventions: Drug: Standard triple therapy
- Bismuth quadruple therapy (Active Comparator): 10 day-bismuth quadruple therapy
  Interventions: Drug: Bismuth quadruple therapy

INTERVENTIONS:
Drug: Standard triple therapy — Lansoprazole 30mg, 2 times a day + Clarithromycin 500mg, 2 times a day + Amoxicillin 1000mg, 2 times a day for 7 days
  Other Names: 7-day PPI-based standard triple therapy
  Arms: Standard triple therapy
Drug: Bismuth quadruple therapy — Lansoprazole 30mg, 2 times a day + Bismuth 300mg, 4 times a day + Tetracycline 500mg, 4 times a day + Metronidazole 500mg, 3 times a day for 10 days
  Other Names: 10-day Bismuth quadruple therapy
  Arms: Bismuth quadruple therapy

SUMMARY:
In this randomized controlled trial, we investigate the effect of 10-day bismuth quadruple therapy in comparison with that of 7-day PPI-based standard triple as 1st line treatment for H. pylori.

DETAILED DESCRIPTION:
Current Helicobacter pylori management guidelines recommend proton-pump inhibitor (PPI)-Clarithromycin containing triple therapy as 1st line treatment. However, in Korea, eradication rates of PPI-Clarithromycin containing triple therapy have been decreased to less than 80% due to increased clarithromycin resistance. In areas of high clarithromycin resistance (resistance rate more than 15%), guidelines recommend bismuth quadruple therapy as a 1st line treatment for H. pylori eradication. Clarithromycin resistance rates reported from 15.7% to 42.1% in Korea, thus, bismuth quadruple therapy may be better 1st line treatment than PPI-Clarithromycin containing triple therapy. However, only one limited study was performed to compare effects of the both treatment regimens in Korea. Thus, studies evaluating the effect of 10-day bismuth quadruple therapy as the first line treatment for H. pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or more including following conditions

  * Family history of gastric cancer
  * Post endoscopic resection status for early gastric cancer or adenoma
  * Peptic ulcer disease (benign gastric ulcer and duodenal ulcer)
  * Chronic gastritis
  * Non-ulcer dyspepsia
  * Healthy adults who want to receive H. pylori treatment
* H. pylori positive by urea breath test, histology, or rapid urease test

Exclusion Criteria:

* History of H. pylori eradication therapy
* History of stomach operation
* Other organ cancer within 5 years
* Liver cirrhosis or Hepatic insufficiency
* Renal insufficiency
* Current treatment for serious medical condition which may hinder participation
* Contraindication or allergy history for H. pylori treatment regimens
* Mental incompetence to understand and sign informed consent
* Incompatible conditions to be included into the trial by investigators' decision
* Inability to provide an informed consent
* History of treatment for peptic ulcer disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-09-28 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | 8 weeks after H. pylori treatment

SECONDARY OUTCOMES:
Complications of H. pylori treatment | 1 month after H. pylori treatment
Compliance to H. pylori treatment | 1 month
H. pylori infection status at 1 year after H. pylori treatment | 1 year after H. pylori treatment
H. pylori reinfection rate | 3 years after success of H. pylori eradication
Factors associated with H. pylori reinfection | 3 years after success of H. pylori treatment

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, M.D., Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim YI, Lee JY, Kim CG, Park B, Park JY, Choi IJ. Ten-day bismuth-containing quadruple therapy versus 7-day proton pump inhibitor-clarithromycin containing triple therapy as first-line empirical therapy for the Helicobacter pylori infection in Korea: a randomized open-label trial. BMC Gastroenterol. 2021 Mar 2;21(1):95. doi: 10.1186/s12876-021-01680-1. PMID 33653284